CLINICAL TRIAL: NCT05190978
Title: Randomized Feasibility Trial for Mesh in Pre-Pectoral Reconstruction
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center (Other); Weill Medical College of Cornell University (Other); Yale University (Other); University of California, Davis (Other); University of Utah (Other); University of California, San Francisco (Other)
Responsible Party: Principal Investigator, Michael R. Delong, Assistant Professor-in-Residence, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 190311
Record Dates: First submitted 2022-01-04; First posted 2022-01-13 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Breast Cancer; Breast Implant; Complications, Infection or Inflammation
Keywords: breast cancer; breast reconstruction; breast implant
MeSH Terms: conditions — Breast Neoplasms; Infections; Inflammation | interventions — Plastic Surgery Procedures

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial
Who Masked: Participant, Outcomes Assessor
Masking Description: Patients will blinded to whether they receive ADM products during their reconstruction.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Acellular Dermal Matrix (Experimental): Patients will receive ADM during their initial tissue expander placement.
  Interventions: Device: Acellular Dermal Matrix
- Control (Active Comparator): Patients will not receive ADM during their initial tissue expander placement.
  Interventions: Procedure: Reconstruction without ADM

INTERVENTIONS:
Device: Acellular Dermal Matrix — Acellular dermal matrix will surgically implanted around the tissue expanders in patients in the ADM cohort.
  Arms: Acellular Dermal Matrix
Procedure: Reconstruction without ADM — Acellular dermal matrix will not be surgically implanted around the tissue expanders in patients in the control cohort.
  Arms: Control

SUMMARY:
Surgical mesh products, particularly acellular dermal matrices (ADM), are now used by the majority of plastic surgeons to assist with the nearly 100,000 prosthetic breast reconstruction procedures in the United States, despite never being approved by Food and Drug Administration (FDA) for this indication. As surgeons transition to placing breast implants above the chest muscle (pre-pectoral), there has been an increasing reliance on these often expensive mesh products without robust evidence to understand their risks and benefits. Our pilot study is a randomized multi-center trial to evaluate surgical mesh assistance in pre-pectoral tissue expander to breast implant reconstruction to address vital questions for women's public health.

DETAILED DESCRIPTION:
One in eight women will develop breast cancer in her lifetime, causing both physical and psychological trauma due to invasive treatments and the distress associated with removal of a breast. Breast reconstruction after mastectomy has become a critical procedure for many women to restore psychological wellbeing, with implant-based reconstruction the most common approach. Nearly 100,000 patients undergo reconstruction with implants every year in the United States.

Surgical mesh devices, particularly acellular dermal matrices, are now used off-label by most reconstructive surgeons performing prosthetic breast reconstruction. In the past decade, surgeons have advocated a transition from submuscular reconstruction (placement of the implant under the pectoralis muscle) to pre-pectoral (placement above the pectoralis) and often consider mesh to be necessary for this procedure. Surgical mesh has not been approved by the FDA for breast reconstruction for either anatomic location. These mesh devices are considered Class III medical devices and FDA recently prioritized the evaluation of these products during a panel meeting in 2019.

No Level I randomized trial has been successfully performed to determine the actual risks and benefits of mesh devices in breast reconstruction. This study proposes a pilot study as the first ever randomized, multi-center trial for mesh assistance in two-stage prosthetic pre-pectoral breast reconstruction, across the major manufacturers. The goals are to demonstrate feasibility of such a study and to generate high level data toward the evaluation of safety and effectiveness of these products for the benefit of women's public health

ELIGIBILITY:
Inclusion Criteria:

* Female patients age 22 to 75 undergoing unilateral or bilateral immediate pre-pectoral reconstruction with tissue expanders
* Prophylactic and oncologic mastectomies are both acceptable
* Nipple sparing and skin sparing mastectomy techniques are both acceptable

Exclusion Criteria:

* Intraoperative assessment demonstrates unfavorable conditions (ie poor mastectomy skin flap thickness or viability) for immediate pre-pectoral reconstruction in any breast
* Bilateral reconstruction patients undergoing contralateral submuscular reconstruction
* Direct-to-implant reconstruction
* Pregnancy
* Delayed reconstruction

Ages: 22 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female patients with breast cancer
Enrollment: 120 (Estimated)
Dates: Start 2022-10-20 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Safety - Major Complications | 2 years
  Relative rate of major complications (requiring unplanned re-admission or re-operation)
Effectiveness - BREASTQ | 2 years
  BREAST-Q validated patient reported questionnaire to assess results of final reconstruction.

SECONDARY OUTCOMES:
Secondary Effectiveness | 2 years
  Time from expander placement to implant exchange
Secondary Safety | 2 years
  Individual complication rates
Capsular Contracture | 2 years
  Rate of capsular contracture

CONTACTS AND LOCATIONS:
Overall Officials: Michael Delong, MD, Principal Investigator — University of California, Los Angeles
Locations (1):
- University of California Los Angeles, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No
All our results will be published in peer-reviewed journals in a timely manner for reference by physicians, manufacturers, regulatory agencies, and patients. As part of the study consent, subjects will be asked whether they agree to share their data in de-identified format with researchers. Data privacy and protection is a top priority. All data made available for public use will be de-identified, i.e., stripped of personally identifiable information (pii) and personal health information (phi) that could be used to deduce the identity of individual subjects, according to the HIPAA Privacy Rule, to comply with the NIH Privacy Rule and Research guidance